CLINICAL TRIAL: NCT05522855
Title: Preliminary Efficacy of a Novel EEG-guided Cognitive Pacing Tool During Concussion Recovery: A Pilot Study
Brief Title: EEG-guided Cognitive Pacing Tool During Concussion Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Matthew Kennedy (Industry)
Responsible Party: Sponsor-Investigator, Dr. Matthew Kennedy, Principal Investigator, Neurovine Inc.
Organization: Neurovine Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV2022-05-002
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Version- EEG Sensorband and mobile application (Experimental): EEG headband to record brain signals. The Sensorband uses Bluetooth to link to the mobile application on a user's device. This raw EEG data is processed on a HIPPA compliant cloud based server and displays mental workload and brain energy data on the application. This can help the user with cognitive pacing to avoid overexertion.
  Interventions: Device: EEG Sensorband and mobile application
- Control Version- EEG Sensorband and mobile application (Active Comparator): EEG headband to record brain signals. The Sensorband uses Bluetooth to link to the mobile application on a user's device. This raw EEG data is processed on a HIPPA compliant cloud based server like the Intervention version, but no mental workload or brain energy data will be displayed.
  Interventions: Device: EEG Sensorband and mobile application

INTERVENTIONS:
Device: EEG Sensorband and mobile application — EEG headband to record brain signals. The Sensorband uses Bluetooth to link to the mobile application on a user's device. This raw EEG data is processed on a HIPPA compliant cloud based server and displays mental workload and brain energy data on the application. This can help the user with cognitive pacing to avoid overexertion. The control version will not display mental workload and brain energy data on the application.

SUMMARY:
This investigation will assess the utility of a novel wearable electroencephalography (EEG) headband linked to a mobile application to monitor cognitive activity post-concussion, and alert a patient when it is time to take a mental break. Personalized cloud-based machine learning algorithms will analyze EEG data in real-time for neural features indicative of mental workload and mental fatigue, and will notify a patient when it is time to rest based on these measures. It is hypothesized that this technology may provide a much needed data-driven management tool to better inform the cognitive pacing process for both patients with concussion, as well as their clinicians.

DETAILED DESCRIPTION:
Despite advancements in the field of concussion care, the individualized nature and nuances of concussion make it a difficult condition to manage. It has been shown that both complete rest or too much activity can prolong recovery from concussion, indicating there is an ideal zone of activity that can aid in concussion recovery. Heart-rate guided sub-symptom aerobic physical activity has been shown to speed concussion recovery and provide an objective measure for patients with concussion to inform their rehabilitative physical activities. However, no such equal exists for guiding cognitive pacing.

This study will utilize a wearable EEG headband linked to a mobile application to monitor cognitive activity post-concussion, and alert a patient when it is time to take a mental break. Personalized cloud-based machine learning algorithms will analyze EEG data in real-time for neural features of mental workload and mental fatigue, and will notify a patient when it is time to rest based on these measures. These algorithms have been developed and validated on healthy participants, and refined in concussion patients in an ongoing observational investigation yet to be published. The proposed investigation is a randomized, prospective pilot study to test the early efficacy of this technology in concussion recovery compared to standard of care alone. The results of this pilot investigation will be used to inform a future large-scale clinical trial to confirm the efficacy of this technology on concussion recovery.

ELIGIBILITY:
Inclusion Criteria: Individuals are eligible to participate if they meet all of the following criteria:

* has been diagnosed with a concussion within previous 6 weeks;
* are between >16 and <55 years of age;
* fluent in English;
* able to attend the baseline testing session within 6 weeks post-injury;
* willing and able to comply with the requirements of the study protocol, including use of intervention;
* able to access a desktop computer or laptop with a colour monitor, reliable internet connection, pointing device,(mouse or trackpad), and modern web browser for administration of ImPACT Version 4.

Exclusion Criteria: Individuals are ineligible to participate if they meet any of the following criteria:

* do not have access to a desktop computer or laptop with the technical requirements to perform ImPACT testing at their home (as described above);
* uncontrolled epilepsy (seizure within 6 months), uncontrolled chronic recurrent migraines, or other neurological disorders that may interfere with concussion recovery and assessment;
* any signs of dementia or other pre-existing cognitive impairment that would prevent them from giving free, informed consent;
* have an implantable electrical device;
* any evidence of the following in addition to concussion diagnosis:

  * documentation that the concussion they had sustained was associated with a Glasgow Coma Scale score ≤ 12 (if available),
  * any findings of trauma on neuroimaging such as brain contusion or hematoma (if available), and
  * any evidence of skull fractures of bony injuries that would require additional rehabilitation.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Immediate Post-Concussion Assessment and Cognitive Testing score | Baseline, post-intervention (2 weeks)
  Change in neurocognitive health and changes in concussion recovery. Higher score indicates improvement.

SECONDARY OUTCOMES:
Study inclusion rate and completion rate to indicate feasibility | Baseline, post-intervention (2 weeks)
  Rates of inclusion, deviations and completion
Rivermead Post-Concussion Symptoms Questionnaire Outcomes | 12 weeks
  Change in symptoms and burden of concussion. Lower score indicates improvement.
Change in Sports Concussion Assessment Tool score | Baseline, post-intervention (2 weeks)
  Change in concussion symptoms. Lower score indicates improvement in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: M Kennedy, Principal Investigator — Neurovine Inc.

IPD SHARING:
Plan to Share IPD: No